CLINICAL TRIAL: NCT05553431
Title: Feasibility of Simplified Permanent Left Bundle Branch Pacing (LBBP) Without Electrophysiological Recording System
Brief Title: Feasibility of Simplified Permanent Left Bundle Branch Pacing Without Electrophysiological Recording System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstWenzhouMU078
Record Dates: First submitted 2022-06-30; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-06

CONDITIONS: Left Bundle Branch Pacing
Keywords: Left Bundle Branch Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No EP system Group (Experimental): Patients were performed left bundle branch pacing without EP system.
  Interventions: Device: Left bundle branch pacing

INTERVENTIONS:
Device: Left bundle branch pacing — Left bundle branch pacing by a CRT device or dual-chamber pacemaker through the pacing lead at left bundle branch region

SUMMARY:
This is a prospective, single-center study of patients with an indication for ventricular pacing who attempted LBBP without electrophysiology recording system (EP system).

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be enrolled into the study. In the study, the implanter was blinded to EP system, only refer to ECG monitoring. The transition of QRS morphology from S-LBBP (or LVSP) to NS-LBBP, abrupt shortening of Stim-LVAT in lead V5, combined with LV septal-derived PVCs and obvious LBB potential in pacing system analyzer were recorded to help the implanter confirm LBB capture. Meanwhile, the technician recorded the data by EP system and evaluated the consistency of the judgment. The primary endpoints included the success rate, procedure-related information, parameters and complications during 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (1) requiring ventricular pacing; (2) older than 18 years; (3) signed informed consent.

Exclusion Criteria:

* (1) acute anterior myocardial infarction; (2) intraventricular conduction delay (IVCD); (3) ventricular septal hypertrophy (end-diastolic thickness over 15 mm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Successful rate | Immediate Postoperative
  Success rate of left bundle branch pacing without EP system
Judgment coincidence rate | Intraoperative
  Coincidence rate between the judgment made by the operator through ECG and PSA with EP system.
Intraoperative complications | Immediate Postoperative
  Intraoperative complications were recorded
Postoperative complications | 3 months
  Postoperative complications were recorded

SECONDARY OUTCOMES:
Procedure duration | Immediate Postoperative
  Total time required for operation
Fluoroscopy time | Immediate Postoperative
  Intraoperative time of radiation use
Change of threshold(V/0.5ms) from immediate postoperative | 3 months
  Threshold for capturing left bundle branch during unipolar pacing
Change of LVEF(%) from baseline | 3 months
  LVEF changes before and after surgery
Change of impedance(Ω) from immediate postoperative | 3 months
  Impedance during unipolar pacing

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Huang, MD, Principal Investigator — Wenzhou 1st Affliated Hopsital, Wenzhou Medical University
Locations (1):
- First Affliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Su L, Wang S, Wu S, Xu L, Huang Z, Chen X, Zheng R, Jiang L, Ellenbogen KA, Whinnett ZI, Huang W. Long-Term Safety and Feasibility of Left Bundle Branch Pacing in a Large Single-Center Study. Circ Arrhythm Electrophysiol. 2021 Feb;14(2):e009261. doi: 10.1161/CIRCEP.120.009261. Epub 2021 Jan 9. PMID 33426907
- [Background] Vijayaraman P, Subzposh FA, Naperkowski A, Panikkath R, John K, Mascarenhas V, Bauch TD, Huang W. Prospective evaluation of feasibility and electrophysiologic and echocardiographic characteristics of left bundle branch area pacing. Heart Rhythm. 2019 Dec;16(12):1774-1782. doi: 10.1016/j.hrthm.2019.05.011. Epub 2019 May 25. PMID 31136869
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611